CLINICAL TRIAL: NCT04579042
Title: Clinical Outcomes After Septoplasty Using Cartilaginous Batten Graft in The Management of The Caudal Septal Deviation
Brief Title: Cartilaginous Batten Graft Septoplasty in Caudal Septal Deviation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelalim, Lecturer of Otorhinolaryngology, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 40-1-2020
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Nasal Septal Deviation
Keywords: Caudal septal deviation; Batten graft; Septoplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septoplasty Using Cartilaginous Batten Graft (Experimental): septoplasty using cartilaginous batten graft in cases with caudal septal deviation
  Interventions: Procedure: cartilaginous batten graft septoplasty

INTERVENTIONS:
Procedure: cartilaginous batten graft septoplasty — septoplasty using cartilaginous batten graft in cases with caudal septal deviation
  Other Names: batten graft septoplasty

SUMMARY:
To evaluate the clinical outcomes of septoplasty using cartilaginous batten graft in cases with caudal septal deviation as regards the relieve of nasal obstruction and aesthetic results.

DETAILED DESCRIPTION:
A prospective study will be conducted over 15 patients indicated for septoplasty.

Preoperative assessment:

History

* NOSE (nasal obstruction septoplasty effectiveness score): Higher NOSE scores indicate worse nasal obstruction (range: 0-100).
* Visual analogue scale (VAS) (0-10) of nasal obstruction:For nasal obstruction

Examination:

* Anterior rhinoscopy: to confirm caudal septal deviation.
* Endoscopic nasal examination: to exclude HIT, polyp, mass and discharge.
* Basal view photograph.
* CT nose and paranasal sinuses to exclude other pathology.

Operative procedures:

* General anesthesia.
* Hemitransfixtion incision on the concave side
* The mucoperichondrial flap of the septum will be elevated
* A contralateral flap will be elevated from the caudal aspect of the cartilage
* Subperichondrial dissection into the nasal floor
* The curved portion of the septal cartilage will be harvested by excision, leaving an L-strut of dorsal and caudal cartilaginous septum
* A caudal septal batten graft created from harvested septal cartilage, then will be sutured using three or four stitches (5-0 polydioxanone sutures).
* If C-shaped caudal deviation without angulation or dislocation, cartilaginous batten graft fixed on the concave side
* If there is angulation of caudal septal end, the caudal strut will be cut by scissors at the most convex point in the caudocephalic direction. Excessive lower and upper caudal struts will be overlapped and sutured together with batten graft
* If dislocated, the septal cartilage will be separated from the anterior nasal spine (ANS) and maxillary crest for reposition. If there is an excessive cartilage portion, it will be removed and then the graft will be sutured
* The hemitransfixion incision will be closed using 5-0 Vicryl
* Internal nasal splint and anterior nasal pack will be placed in both sides

ELIGIBILITY:
Inclusion Criteria:

- Patient presented with nasal obstruction or disfigurement due to anterocaudal septal deviation.

Exclusion Criteria:

* Previous septal surgery
* Deformed nose, which necessitate external rhinoplasty approach.
* Other endonasal cause of nasal obstruction other than deviated nasal septum
* Bleeding disorder or systemic diseases.
* Patient who will not complete the follow up periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Nasal obstruction | 3 months
  We will use the validated Nasal obstruction septoplasty effectiveness score: (range: 0-100) Higher NOSE scores indicate worse nasal obstruction.

SECONDARY OUTCOMES:
Aesthetic results | 6 months
  Basal view photography:
  Two independent observers will review the photographs and 4-point grading system will be used to evaluate results:
  * Grade I: Will indicate that the patient has little or no photographic evidence of residual caudal septal deviation.
  * Grade II: The caudal septal deviation show marked improvement but still detectable by careful observation.
  * Grade III: The caudal deviation is only mildly improved or not improved from the preoperative assessment.
  * Grade IV: The caudal deviation is worse after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman A Abdelalim, MD, Principal Investigator — Benha University; Ashraf S El-Hamshary, MD, Study Chair — Benha University; Ibrahim S Reyad, Resident, Study Chair — Benha University
Locations (1):
- Benha University Hospital, Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910
- [Background] Chung YS, Seol JH, Choi JM, Shin DH, Kim YW, Cho JH, Kim JK. How to resolve the caudal septal deviation? Clinical outcomes after septoplasty with bony batten grafting. Laryngoscope. 2014 Aug;124(8):1771-6. doi: 10.1002/lary.24491. Epub 2013 Dec 9. PMID 24323627